CLINICAL TRIAL: NCT00987272
Title: A Phase III Study of Olopatadine HCl Ophthalmic Solutions Compared to Vehicle Using the CAC Model of Acute Allergic Conjunctivitis in Japanese Subjects
Brief Title: Study of Olopatadine HCl Ophthalmic Solutions Compared to Vehicle Using the Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-09-044
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergies; Ocular
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pataday+Pataday Vehicle (Experimental): Olopatadine Hydrochloride Ophthalmic Solution 0.2%, 1 drop in 1 eye and Olopatadine 0.2% Vehicle in the contralateral eye
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%; Drug: Olopatadine 0.2% Vehicle
- Patanol+Patanol Vehicle (Active Comparator): Olopatadine Hydrochloride Ophthalmic Solution, 0.1%, 1 drop in 1 eye and Olopatadine 0.1% Vehicle in the contralateral eye
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.1%; Drug: Olopatadine 0.1% Vehicle

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%
  Other Names: PATADAY®
  Arms: Pataday+Pataday Vehicle
Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.1%
  Other Names: PATANOL®
  Arms: Patanol+Patanol Vehicle
Drug: Olopatadine 0.2% Vehicle — Inactive ingredients used as placebo comparator
  Arms: Pataday+Pataday Vehicle
Drug: Olopatadine 0.1% Vehicle — Inactive ingredients used as placebo comparator
  Arms: Patanol+Patanol Vehicle

SUMMARY:
The purpose of the study is to demonstrate safety and efficacy of Olopatadine 0.2% compared to its vehicle in Japanese subjects in the treatment of acute allergen-mediated conjunctivitis using the conjunctival allergen challenge (CAC) test.

ELIGIBILITY:
Inclusion Criteria:

* Japanese ethnicity.
* Seasonal Allergic Conjunctivitis--asymptomatic.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Manifest signs and symptoms of clinically active allergic conjunctivitis in either eye (>1 for redness in any of the 3 vessels beds - conjunctival, episcleral, ciliary - or itching >0) at the start of any visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Mean Ocular Itching Score | Day 0 of treatment: 3, 5, and 10 minutes post CAC

SECONDARY OUTCOMES:
Mean Total Redness Score | Day 0 of treatment: 3, 10, 20 minutes post-CAC

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Smith, BS, Study Director — Alcon Research